CLINICAL TRIAL: NCT06332105
Title: The Effects of an Innovative Glycomacropeptide Based Protein Supplement Purified to Lower the Phenylalanine Content for the Treatment of Paediatric Patients With Phenylketonuria
Brief Title: Evaluation of Low Phenylalanine Formulas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ajinomoto Co., Inc. (Industry)
Collaborators: Birmingham Children's Hospital (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CUK001
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: 2-stage, 15-week randomized crossover trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB: GMP-AA -> L-AA (Active Comparator): After an initial washout period of 2 weeks, participants randomised to Sequence AB will consume GMP-AA for 3 months whilst keeping a food diary and sending blood spots for twice weekly analysis. At the end of 3 months there is a further 2 week washout period with L-AA, after which the participant will consume L-AA for 3 months whilst keeping a food diary and sending blood spots for twice weekly analysis.
  Interventions: Dietary Supplement: Glytactin
- Sequence BA: L-AA -> GMP-AA (Placebo Comparator): After an initial washout period of 2 weeks, participants randomised to Sequence BA will consume L-AA for 3 months whilst keeping a food diary and sending blood spots for twice weekly analysis. At the end of 3 months there is a further 2 week washout period with L-AA, after which the participant will consume GMP-AA for 3 months whilst keeping a food diary and sending blood spots for twice weekly analysis.
  Interventions: Dietary Supplement: L-AA

INTERVENTIONS:
Dietary Supplement: Glytactin — Glycomacropeptide based protein substitute for dietary treatment of PKU
  Other Names: Glytactin Build 20 Flavours; Glytactin Ready To Drink (RTD) 15 Lite; Glytactin Build 10
  Arms: Sequence AB: GMP-AA -> L-AA
Dietary Supplement: L-AA — Amino acid based protein substitute for dietary treatment of PKU
  Arms: Sequence BA: L-AA -> GMP-AA

SUMMARY:
Ajinomoto Cambrooke has developed a PKU protein substitute that is a proprietary blend of purified Glycomacropeptide (GMP) and essential amino acids, under the brand name Glytactin®. One serving of such Glytactin® products contains 20mg or less of Phenylalanine (Phe). The aim of the proposed study is to use this purified GMP-AA-based protein substitute, with less Phe per gram of protein equivalent than other commercially available products, in children with PKU at 100% of their protein substitute intake and evaluate its efficacy and the change in blood Phe in comparison to Phe-free L-AA-based protein substitutes.

DETAILED DESCRIPTION:
Study Design This is a 2-stage, 15-week randomized crossover trial. The randomized crossover design was chosen as it reduces the influence of differences among individuals; and it offers statistical efficiency (requires fewer subjects than non-crossover designs).

In summary, 2 groups of 9 participants each will be assigned to either (1) sequence 1: take GMP-AA-based PS for the first 4 weeks and then take only L-AA-based Protein Substitute for 4 weeks, or (2) take only L-AA-based Protein Substitute for the first 4 weeks and then take GMP-AA-based PS for 4 weeks. At the end of the first 4 weeks, a 2-week washout period will follow with both groups only consuming L-AA-based PS. Randomization will be generated by a block randomization system and the random order will be kept within a sealed envelope.

Primary research objective The principal research objective of this study is to evaluate the effect on Phe levels of a low-Phe diet combined with a purified GMP-AA-based protein substitute (containing 1 mg Phe/g Protein Equivalent), in the treatment of paediatric patients with PKU.

Secondary research objectives The secondary objectives of the study aim to investigate whether there are any differences between the GMP-AA-based protein substitute and L-AA-based protein Substitute in the frequency and quantity of protein substitute intake, if any GI (gastrointestinal) symptoms occur with ingestion of the GMP-AA-based protein substitute, effect on satiety (hunger) and mood and any differences in anthropometric data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PKU, aged 5 to 16 years of age, currently compliant with protein restricted diet and L-AA- and/or GMP-AA-based protein substitute willing to switch to a GMP-AA-based only product for 4 weeks.

  * 2 out of 4 last blood Phe levels within target range (i.e. 50%): Target range 120-360µmol/l <12 years Target range 120-600µmol/l >12 years

Exclusion Criteria:

* • Milk protein allergy

  * Pregnancy
  * Severe medical diagnosis not related to PKU
  * Treatment with Sapropterin hydrochloride (KUVAN)

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in blood Phe in | 16 weeks
  Change in blood Phe in subjects ingesting purified GMP-AA-protein substitute compared with the change when ingesting L-AA-protein substitute

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, BSc PhD, Principal Investigator — Birmingham Women and Children's Hospital
Locations (2):
- United Kingdom (2):
  - Birmingham Women and Children's Hospital, Birmingham, West Midlands
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No